CLINICAL TRIAL: NCT04089618
Title: Meditation Based Lifestyle Modification in Chronic Pain
Acronym: MBLM-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonie Kliniken Zschadraß (Other)
Collaborators: Chemnitz University of Technology (Other); Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Holger C. Bringmann, Principal investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBLM-P
Record Dates: First submitted 2019-09-07; First posted 2019-09-13 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Pain, Chronic
Keywords: Yoga; Meditation; Yoga Philosophy; Mantra; Mind-Body
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Single Case Research (SCR), also known as single case experimenal design (SCED). This is a reserach methodology using a single unit of analysis and characterized by repeated measures over time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline 10 Days (Experimental): 10 days baseline before intervention starts.
  Interventions: Behavioral: MBLM
- Baseline 17 Days (Experimental): 17 days baseline before intervention starts.
  Interventions: Behavioral: MBLM
- Baseline 24 Days (Experimental): 24 days baseline before intervention starts.
  Interventions: Behavioral: MBLM

INTERVENTIONS:
Behavioral: MBLM — Complex 8 week Mind-Body program.

SUMMARY:
MBLM is a holistic therapy for people with mental disorders whose feasibility positive effects on patients with depression have already been demonstrated in clinical application and a piloted study. In the present trial, the feasibility and effect of MBLM on patients with chronic pain will be investigated.

DETAILED DESCRIPTION:
MBLM expands existing concepts of mind-body medicine with ethical and spiritual concepts from the traditional Patanjali Yoga system, which can act as a coping factor on the one hand, and higher motivation and deepening of self-administered practice (mindfulness based exercises, body-oriented yoga exercises and mantra meditation). MBLM aims to establish an exercise routine in the daily lives of the participants, which leads to salutogenesis. The promotion of mental health through meditation and yoga has been well documented, also in clinical populations. The effects of meditation and yoga on addiction and pain are promising, but there is still a need for research. Furthermore, the preventive potential of the MBLM program will be examined for healthy volunteers, analogous to the already well-researched and widely used MBSR (Mindfulness Based Stress Reduction) program, which was originally also developed for patients with pain disorders.

The study will be conducted as an experimental single case analysis with multiple baseline design. Randomization takes place over time instead of control groups.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients
2. Current diagnosis of a chronic pain disorder.
3. Over 18 years old.
4. Physically able to perform simple yoga postures and sit for 20 minutes.
5. Have given your written consent to participate in the study.

Exclusion Criteria:

1. Psychotic symptoms
2. Acute suicidality
3. obsessive-compulsive disorder
4. Cerebro-organic diseases with clinically relevant symptoms
5. Severe multimorbidity
6. Current participation in another meditation or yoga study
7. Regular meditation or yoga practice (> once a week in the last 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Pain VAS | through study completion, daily for around 3 months
  Visual Analog Scale for Pain
Pain medication | through study completion, daily for around 3 months
  Use of pain medication
Well-Being | through study completion, daily for around 3 months
  The WHO-5 Well-Being Scale (WHO-5; World Health Organisation, 1998)

SECONDARY OUTCOMES:
Emotion Regulation | through study completion, weekly for around 3 months
  Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2003)
Body awareness | through study completion, twice weekly for around 3 months
  adapted from Private-Body-Consciousness-Scale (PBCS; Miller, Murphy, & Buss, 1981), Body-Awareness-Questionnaire" (BAQ; Shields, Mallory & Simon, 1989) and Multidimensional Assessment of Interoceptive Awareness" (MAIA; Mehling et al., 2012)
Mind-Wandering | through study completion, weekly for around 3 months
  a) Mind-Wandering Questionnaire (MWQ; Mrazek, Phillips, Franklin, Broadway, & Schooler, 2013)
Depression, Anxiety & Stress | through study completion, weekly for around 3 months
  DASS (Nilges & Essau, 2015)
Pain Self Efficacy | through study completion, weekly for around 3 months
  PAIN SELF EFFICACY QUESTIONNAIRE (PSEQ) M.K.Nicholas (1989)

OTHER OUTCOMES:
Quality of Life | at week 0 and week 11
  WHOQol-BREF
Chronic Pain Self-Efficacy | at week 0 and week 11
  CPSS (Anderson et al, 1995)
Distress Tolerance | at week 0 and week 11
  Distress tolerance (Simons & Gaher, 2005)
Spiritual and Religious Attitudes in Dealing with Illness | at week 0 and week 11
  SpREUK (Büssing A., 2010)
Trigunas - Emotion, Cognition and Health Behaviour | at week 0 and week 11
  TGS Subscales (Puta & Sedlmeier, 2014)
Illness Cognition | at week 0 and week 11
  Illness Cognition Questionnaire for Chronic Diseases (Evers et al., 2001)

CONTACTS AND LOCATIONS:
Locations (1):
- Diakoniekliniken Zschadraß, Colditz, Saxony, Germany